CLINICAL TRIAL: NCT02830594
Title: Combining Pembrolizumab and Palliative Radiotherapy in Gastroesophageal Cancer to Enhance Anti-Tumor T Cell Response and Augment the Abscopal Effect
Brief Title: Pembrolizumab and Palliative Radiation Therapy in Treating Patients With Metastatic Esophagus, Stomach, or Gastroesophageal Junction Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16099; NCI-2016-00686 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 16099 (Other: City of Hope Medical Center)
Record Dates: First submitted 2016-05-18; First posted 2016-07-13 (Estimated); Results first posted 2022-06-30 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Gastric Adenocarcinoma; Gastric Squamous Cell Carcinoma; Gastroesophageal Junction Adenocarcinoma; Metastatic Malignant Neoplasm in the Stomach; Stage IV Esophageal Adenocarcinoma AJCC v7; Stage IV Esophageal Squamous Cell Carcinoma AJCC v7
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma | interventions — Radiation; pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (pembrolizumab, RT) (Experimental): INITIAL TREATMENT: Patients undergo palliative external beam RT daily. On day 1, patients undergo the first RT fraction and then receive pembrolizumab intravenously (IV) over 30 minutes. Cycles repeat every 3 weeks for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  SECOND PHASE: Patients who achieve a complete response, stop study treatment, and then experience radiographic disease progression may be eligible for the second phase at the discretion of the investigator if no cancer treatment was administered since the last dose of pembrolizumab and trial eligibility safety parameters are met. Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 17 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Radiation: External Beam Radiation Therapy; Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Radiation: External Beam Radiation Therapy — Undergo palliative external beam radiation therapy
  Other Names: Definitive Radiation Therapy; EBRT; External Beam Radiation; External Beam Radiotherapy; External Beam RT; external radiation; External Radiation Therapy; external-beam radiation; Radiation, External Beam
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab and palliative radiation therapy works in treating patients with esophagus, stomach, or gastroesophageal junction cancer that has spread to other parts of the body. Monoclonal antibodies, such as pembrolizumab, may interfere with the ability of tumor cells to grow and spread. Palliative radiation therapy, such as external beam radiation therapy, uses high energy beams to treat symptoms that are caused by tumors. Giving pembrolizumab together with palliative radiation therapy may work better in treating patients with esophagus, stomach, or gastroesophageal junction cancer that has spread to other parts of the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish that the combination of pembrolizumab and traditional external beam multifractionated radiation therapy (RT) to the primary tumor or a single target metastatic site of patients with metastatic gastric, esophageal, and/or gastroesophageal junction (GEJ) cancers will lead to an increase in tumor infiltrating cytotoxic T-cells and circulating cytotoxic T cells and a reduction in immunosuppressive regulatory T cells (Tregs) and myeloid-derived suppressor cells (MDSCs) in metastatic sites.

SECONDARY OBJECTIVES:

I. To establish that the combination of pembrolizumab and RT is feasible in the patient population and evaluate toxicities per National Cancer Institute (NCI) Common Toxicity Criteria for Adverse Events (CTCAE) version (ver.) 4.03.

II. To evaluate overall response rate (ORR) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune related (ir)RECIST in this treatment population and correlate with tumor T-cell response.

III. To evaluate progression-free (PFS) and overall survival (OS) in this treatment population.

EXPLORATORY OBJECTIVES:

I. To measure changes in whole genome serum micro ribonucleic acid (miRNA) signature before and after protocol therapy and correlate with tumor/immune/stromal cell miRNA expression profiling determined by deep sequencing.

II. To measures changes in fecal and oral microbiomic diversity and correlative with ORR, PFS, and OS.

III. To assess germline mutations in a panel of miRNA regulatory genes using the MiraDx assay as predictors of response and toxicity to pembrolizumab and RT.

OUTLINE:

INITIAL TREATMENT: Patients undergo palliative external beam RT daily. On day 1, patients undergo the first RT fraction and then receive pembrolizumab intravenously (IV) over 30 minutes. Cycles repeat every 3 weeks for up to 35 cycles in the absence of disease progression or unacceptable toxicity.

SECOND PHASE: Patients who achieve a complete response, stop study treatment, and then experience radiographic disease progression may be eligible for the second phase at the discretion of the investigator if no cancer treatment was administered since the last dose of pembrolizumab and trial eligibility safety parameters are met. Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 17 cycles in the absence of disease progression or unacceptable toxicity.

After completion of treatment, patients are followed up at 30 days, every 6 weeks for 1 year, and then every 9 and 12 weeks for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Documented informed consent of the participant
* Willing to provide tumor tissue amenable to ultrasound or computed tomography (CT)-guided biopsy for biomarker analyses

  * Patients with malignant ascites are permitted to participate and provide ascites samples for biomarker analyses
  * Patents receiving radiation to a single metastatic site in which only the primary tumor is accessible for biopsy by endoscopy will also be eligible
* Eastern Cooperative Oncology Group (ECOG) performance status of =< 1
* Life expectancy of >= 3 months
* Diagnosis of metastatic squamous cell carcinoma and/or adenocarcinoma of the esophagus, gastroesophageal junction, or stomach in need of palliative radiotherapy to the primary tumor or a single metastatic site for symptoms such as pain, dysphagia, and/or gastrointestinal bleeding

  * Patients with adenocarcinoma histology and known human epidermal growth factor receptor 2 (HER2) overexpressing disease are permitted to participate if the progressed or are intolerant of prior trastuzumab-containing therapy
* Measurable metastatic sites of disease outside of the target lesion undergoing palliative radiation based on RECIST 1.1 as assessed by the investigator
* Have no limits on prior lines of therapy or may be treatment-naive if in need of palliative RT provided the patient has not received prior anti-programmed cell death protein 1(PD-1), anti-programmed cell death 1 ligand 1 (PD-L1), or anti-programmed cell death 1 ligand 2 (PD-L2) therapy
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelets >= 100,000/mm^3
* Hemoglobin >= 9 g/dL

  * May receive transfusion to meet this goal
* Total serum bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN if total bilirubin levels > 1.5 x ULN
* Albumin >= 2.5 mg/dL
* Aspartate aminotransaminase (AST) and alanine aminotransferase (ALT) =< 2.5 x ULN OR =< 5.0 x ULN if liver metastases present
* Serum creatinine =< 1.5 x ULN OR creatinine clearance (if measured or calculated per institutional standard) >= 60 mL/min if creatinine levels > 1.5 x ULN

  * Glomerular filtration rate (GFR) can also be used in place of creatinine or creatinine clearance (CrCl)
* If not receiving anticoagulants: international normalized ratio (INR) OR prothrombin (PT) =< 1.5 x ULN; if on anticoagulant therapy: PT must be within therapeutic range of intended use of anticoagulants
* If not receiving anticoagulants: activated partial thromboplastin time (aPTT) =< 1.5 x ULN; if on anticoagulant therapy: aPTT must be within therapeutic range of intended use of anticoagulants
* Negative urine or serum pregnancy test (female of childbearing potential only)

  * If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
* Female of childbearing potential: willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication

  * Childbearing potential defined as not being surgically sterilized or have not been free from menses for > 1 year
* Male: use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy

Exclusion Criteria:

* Anti-PD-1, anti-PD-L1, or anti-PD-L2 agents
* Prior radiation therapy within the field of the target lesion that in the opinion of the treating radiation oncologist would preclude further palliative radiation to a dose of 30 gray (Gy)
* Anti-cancer monoclonal antibody (mAb) within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier
* Chemotherapy, targeted small molecule therapy, or radiation therapy within 2 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from adverse events due to a previously administered agent

  * Note: Subjects with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Live vaccine within 30 days of planned start of study therapy

  * Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are live attenuated vaccines, and are not allowed
* Immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Investigational device within 4 weeks of the first dose of treatment
* Currently receiving an investigational agent
* About to undergo palliative radiation for a symptomatic central nervous system (CNS) metastasis
* Systemic steroid therapy
* Hypersensitivity to pembrolizumab or any of its excipients
* Diagnosis of immunodeficiency
* Active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease modifying agents, corticosteroids or immunosuppressive drugs)

  * Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment
* Known history of, or any evidence of active, non-infectious pneumonitis
* Current active infection requiring systemic therapy
* Known history of active tuberculosis (TB), human immunodeficiency virus (HIV) 1/2, hepatitis B or hepatitis C
* Known additional malignancy that is progressing or requires active treatment

  * Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis

  * Subjects with previously treated brain metastases may participate provided they are stable, have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment; this exception does not include carcinomatous meningitis which is excluded regardless of clinical stability
* History or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Pregnant or breastfeeding (female only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-10-05 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2024-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marwan Fakih, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope Medical Center, Duarte, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Pembrolizumab, RT): INITIAL TREATMENT: Patients undergo palliative external beam RT daily. On day 1, patients undergo the first RT fraction and then receive pembrolizumab intravenously (IV) over 30 minutes. Cycles repeat every 3 weeks for up to 35 cycles in the absence of disease progression or unacceptable toxicity.
  SECOND PHASE: Patients who achieve a complete response, stop study treatment, and then experience radiographic disease progression may be eligible for the second phase at the discretion of the investigator if no cancer treatment was administered since the last dose of pembrolizumab and trial eligibility safety parameters are met. Patients receive pembrolizumab IV over 30 minutes on day 1. Cycles repeat every 3 weeks for up to 17 cycles in the absence of disease progression or unacceptable toxicity.
  External Beam Radiation Therapy: Undergo palliative external beam radiation therapy
  Laboratory Biomarker Analysis: Correlative studies
  Pembrolizumab: Given IV
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab, RT)
Started | 14
Completed | 14
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab, RT)
Number analyzed (Participants) | 14
Age, Continuous [Median (Full Range); unit: years] | 67 [40 to 91]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 7
  Asian | 5
  African American | 1
  Hispanic | 1
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Changes in Combined Positive Scoring (CPS) in Non-irradiated Sites Assessed by Flow Cytometry
Description: Multicolor immunofluorescence was performed to quantitate analogous CPS expression in pre- and posttreatment biopsies. Difference in MIDS expression between pre- and posttreatment was tested using a Paired T-test.
Time Frame: Baseline to 105 weeks
Population: One patient did not undergo any biopsies due to site of metastasis not being visualized under image guidance and 2 patients did not undergo the second biopsy for patient safety. Four patients had posttreatment biopsies without any viable cancer cells but only residual stromal tissue.
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Treatment (Pembrolizumab, RT)
Number analyzed (Participants) | 7
fold change | 3.9 (7.0)
Statistical Analysis 1: Comparison: Treatment (Pembrolizumab, RT); Test type: Equivalence — Specifically, a sample-size of 14 patients will have 80% power to detect an effect size of 0.71 using a paired t-test with a 0.05 one-sided significance level. The effect size is the mean difference divided by the standard deviation of the difference; p = 0.60, Paired t Test

2. Primary Outcome: Changes in Tumor Proportion Scores (TPS) in Non-irradiated Sites Assessed by Flow Cytometry
Description: Multicolor immunofluorescence was performed to quantitate analogous TPS expression in pre- and posttreatment biopsies. Difference in MIDS expression between pre- and posttreatment was tested using a Paired T-test.
Time Frame: Baseline to 105 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Treatment (Pembrolizumab, RT)
Number analyzed (Participants) | 7
fold change | 0.3 (1.7)
Statistical Analysis 1: Comparison: Treatment (Pembrolizumab, RT); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.87, Paired t Test

3. Primary Outcome: Changes in Myeloid-derived Suppressor Cells (MDSC) in Non-irradiated Sites Assessed by Flow Cytometry
Description: Multicolor immunofluorescence was performed to quantitate analogous MIDS expression in pre- and posttreatment biopsies. Difference in MIDS expression between pre- and posttreatment was tested using a Paired T-test.
Time Frame: Baseline to 105 weeks
Population: as for outcome 1
Measure: Mean (Standard Error); unit: fold change
Arm/Group | Treatment (Pembrolizumab, RT)
Number analyzed (Participants) | 7
fold change | 3.6 (7.2)
Statistical Analysis 1: Comparison: Treatment (Pembrolizumab, RT); Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p = 0.64, Paired t Test

4. Secondary Outcome: Incidence of Treatment Related Adverse Events of Pembrolizumab
Description: Graded per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03. Adverse events with incidence greater than 10%. An adverse event is any untoward medical experience or change of an existing condition that occurs during or after treatment, whether or not it is considered to be related to the protocol intervention. Serious Adverse Events as: Death; Is life-threatening experience (places the subject at immediate risk of death from the event as it occurred); Unplanned hospitalization (equal to or greater than 24 hours) or prolongation of existing hospitalization; A persistent or significant disability/incapacity; A congenital anomaly/birth defect; Secondary malignancy; Any other adverse event that, based upon appropriate medical judgment, may jeopardize the subject's health and may require medical or surgical intervention to prevent one of the outcomes listed above.
Time Frame: Up to 36 months
Measure: Number; unit: participants
Arm/Group | Treatment (Pembrolizumab, RT)
Number analyzed (Participants) | 14
participants
  Grade 1-2 Fatigue | 4
  Grade 1-2 Pruritus | 4
  Grade 1-2 Pneumonitis | 2
  Grade 1-2 Skin Rash | 2
  Grade 1-2 Constipation | 2
  Grade 1-2 Xerostomia | 2
  Grade 1-2 Thrombocytopenia | 2
  Grade 3-4 Diarrhea | 1
  Grade 3-4 Enterocolitis | 1

5. Secondary Outcome: Overall Response Rate (ORR)
Description: Response was assessed using Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 and immune related (ir)RECIST. Overall Response (OR) = CR + PR.
Time Frame: Up to 36 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pembrolizumab, RT)
Number analyzed (Participants) | 14
percentage of participants | 28.6 [8.4 to 58.1]

6. Secondary Outcome: Progression-free Survival (PFS)
Description: Estimated using the product-limit method of Kaplan and Meier. Event defined as progression or death from any cause. Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions. irPD defined as a minimum 20% increase and minimum 5 mm absolute increase in TMTB compared to nadir, or irPD for non-target or new non-measurable lesions. Confirmation of progression is recommended minimum 4 weeks after the first irPD assessment.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pembrolizumab, RT)
Number analyzed (Participants) | 14
Months | 1.3 [1.1 to NA] — NA - The upper limit of the 95% confidence interval was not calculable because an insufficient number of participants reached the event at the final time point for assessment.

7. Secondary Outcome: Overall Survival (OS)
Description: Estimated using the product-limit method of Kaplan and Meier. Event defined as death from any cause.
Time Frame: Up to 36 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Treatment (Pembrolizumab, RT)
Number analyzed (Participants) | 14
Months | 3.7 [2.0 to 26.2]

ADVERSE EVENTS:
Time Frame: Adverse events occurred over a period of 41 months.
Description: "Other Adverse Events" include all events that were not severe adverse events regardless of grade or relation to treatment.
Arm/Group | Treatment (Pembrolizumab, RT)
All-Cause Mortality (participants affected / at risk) | 9/14
Serious Adverse Events (participants affected / at risk) | 9/14
Other Adverse Events (participants affected / at risk) | 14/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, RT) (N=14)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Pericardial effusion (Cardiac disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Enterocolitis (Gastrointestinal disorders) | 1 (1)
Lung infection (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pembrolizumab, RT) (N=14)
Anemia (Blood and lymphatic system disorders) | 5 (34)
Blood and lymphatic system disorders - O (Blood and lymphatic system disorders) | 1 (2)
Cardiac disorders - Other, specify (Cardiac disorders) | 1 (6)
Pericardial effusion (Cardiac disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 4 (7)
Diarrhea (Gastrointestinal disorders) | 2 (27)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Dysphagia (Gastrointestinal disorders) | 2 (8)
Esophagitis (Gastrointestinal disorders) | 1 (1)
Flatulence (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 1 (2)
Nausea (Gastrointestinal disorders) | 5 (6)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (3)
Edema limbs (General disorders) | 2 (3)
Fatigue (General disorders) | 8 (23)
Fever (General disorders) | 1 (1)
Infusion related reaction (General disorders) | 1 (1)
Non-cardiac chest pain (General disorders) | 1 (1)
Pain (General disorders) | 1 (3)
Infections and infestations - Other, spe (Infections and infestations) | 2 (2)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 3 (6)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Blood bilirubin increased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 1 (18)
Platelet count decreased (Investigations) | 2 (11)
White blood cell decreased (Investigations) | 1 (16)
Anorexia (Metabolism and nutrition disorders) | 3 (4)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (2)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 8 (16)
Hypocalcemia (Metabolism and nutrition disorders) | 4 (6)
Hypokalemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 8 (18)
Hypophosphatemia (Metabolism and nutrition disorders) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (13)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Musculoskeletal and connective tissue di (Musculoskeletal and connective tissue disorders) | 2 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (2)
Dysphasia (Nervous system disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Nervous system disorders - Other, specif (Nervous system disorders) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (36)
Confusion (Psychiatric disorders) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (23)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 4 (13)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (18)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (2)
Skin and subcutaneous tissue disorders - (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (11)
Hypotension (Vascular disorders) | 2 (24)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-10-16): https://cdn.clinicaltrials.gov/large-docs/94/NCT02830594/Prot_SAP_000.pdf
  • Informed Consent Form (2017-09-06): https://cdn.clinicaltrials.gov/large-docs/94/NCT02830594/ICF_001.pdf